CLINICAL TRIAL: NCT02970942
Title: This Trial is Conducted Globally. The Aim of This Trial is to Investigate Efficacy and Safety of Three Dose Levels of Subcutaneous Semaglutide Once Daily Versus Placebo in Subjects With Non-alcoholic Steatohepatitis
Brief Title: Investigation of Efficacy and Safety of Three Dose Levels of Subcutaneous Semaglutide Once Daily Versus Placebo in Subjects With Non-alcoholic Steatohepatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9931-4296; 2016-000685-39 (EudraCT Number); U1111-1179-7464 (Other: WHO)
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Hepatobiliary Disorders; Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Digestive System Diseases; Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Semaglutide 0,1 mg (Experimental)
  Interventions: Drug: Semaglutide
- Semaglutide 0,2 mg (Experimental)
  Interventions: Drug: Semaglutide
- Semaglutide 0,4 mg (Experimental)
  Interventions: Drug: Semaglutide
- Placebo 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Once daily administration of semaglutide subcutaneously (s.c., under the skin) in three different doses (0.1 mg, 0.2 mg and 0.4 mg)
  Arms: Semaglutide 0,1 mg; Semaglutide 0,2 mg; Semaglutide 0,4 mg
Drug: Placebo — Once daily administration subcutaneously ( s.c., under the skin)
  Arms: Placebo 1; Placebo 2; Placebo 3

SUMMARY:
Investigation of efficacy and safety of three dose levels of subcutaneous semaglutide once daily versus placebo in subjects with non-alcoholic steatohepatitis

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial except for protocol described pre-screening activities which require a separate informed consent. - Male or female, aged 18-75 years (both inclusive) (for Japan: male or female aged 20-75 years (both inclusive)) at the time of signing informed consent - Local histological diagnosis of NASH followed by histological confirmation of NASH based on central pathologist evaluation of a liver biopsy obtained up to 21 weeks before screening - Histologic evidence of NASH based on central pathologist evaluation of a liver biopsy obtained up to 21 weeks before screening. - NASH fibrosis stage 1, 2 or 3 according to the NASH CRN fibrosis staging system based on central pathologist evaluation Exclusion Criteria: - Known or suspected abuse of alcohol (above 20 g/day for women or above 30 g/day for men), alcohol dependence* or narcotics. (* = assessed by the Alcohol Use Disorders Identification Test (AUDIT questionnaire)) - Diagnosis of type 1 diabetes according to medical records - HbA1c above 10% at screening - History or presence of pancreatitis (acute or chronic) - Calcitonin equal or above 50 ng/L at screening - Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma. Family is defined as a first degree relative - Body Mass Index (BMI) ≤ 25.0 kg/sqm at the screening visit (visit 1) - Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (130):
- United States (35):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Coronado, California
  - Novo Nordisk Investigational Site, Costa Mesa, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Panorama City, California
  - Novo Nordisk Investigational Site, Rialto, California
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lakewood Rch, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocoee, Florida
  - Novo Nordisk Investigational Site, Sarasota, Florida
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Rochester, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Manhasset, New York
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Hermitage, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Rollingwood, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Burlington, Vermont
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington
- Australia (5):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Kingswood, New South Wales
  - Novo Nordisk Investigational Site, Westmead, New South Wales
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Fitzroy, Victoria
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Belgium (3):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Canada (8):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Denmark (2):
  - Novo Nordisk Investigational Site, Aarhus N
  - Novo Nordisk Investigational Site, Hvidovre
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (10):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Clermont-Ferrand
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pessac
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Vénissieux
- Greece (4):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Goudi, Athens
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Thessaloniki
- Japan (14):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Fukui-shi, Fukui
  - Novo Nordisk Investigational Site, Kamigyo-ku, Kyoto
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Nagakute-shi, Aichi
  - Novo Nordisk Investigational Site, Nara-shi, Nara
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hyogo
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Otsu-shi, Shiga
  - Novo Nordisk Investigational Site, Saga-shi, Saga
  - Novo Nordisk Investigational Site, Shimonoseki-shi, Yamaguchi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Takamatsu-shi, Kagawa
  - Novo Nordisk Investigational Site, Toyoake-shi, Aichi
- Netherlands (8):
  - Novo Nordisk Investigational Site, Alkmaar
  - Novo Nordisk Investigational Site, Amstelveen
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Maastricht
  - Novo Nordisk Investigational Site, Nijmegen
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (13):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Kemerovo
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ulyanovsk
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Spain (6):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Majadahonda
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- United Kingdom (13):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Portsmouth
  - Novo Nordisk Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
According to Novo Nordisk disclosure commitment on novonordisk.com

REFERENCES:
- [Result] Newsome PN, Buchholtz K, Cusi K, Linder M, Okanoue T, Ratziu V, Sanyal AJ, Sejling AS, Harrison SA; NN9931-4296 Investigators. A Placebo-Controlled Trial of Subcutaneous Semaglutide in Nonalcoholic Steatohepatitis. N Engl J Med. 2021 Mar 25;384(12):1113-1124. doi: 10.1056/NEJMoa2028395. Epub 2020 Nov 13. PMID 33185364
- [Derived] Nitze LM, Ratziu V, Sanyal AJ, Wong VW, Balendran C, Fleckner J, Skalshoi Kjaer M, Krarup N, Anstee QM. Exploration of Multiple Non-Invasive Tests for Assessing Response to Treatment in a Semaglutide Phase 2b Trial in Patients with MASH. Aliment Pharmacol Ther. 2026 Feb;63(3):396-404. doi: 10.1111/apt.70376. Epub 2025 Sep 23. PMID 40985232
- [Derived] Schattenberg JM, Gronbaek H, Kliers I, Ladelund S, Long MT, Nygard SB, Sanyal AJ, Davies MJ. Proteomic signatures reflect effects of semaglutide treatment for MASH. JHEP Rep. 2025 Jul 22;7(10):101521. doi: 10.1016/j.jhepr.2025.101521. eCollection 2025 Oct. PMID 40980163
- [Derived] Ratziu V, Francque S, Behling CA, Cejvanovic V, Cortez-Pinto H, Iyer JS, Krarup N, Le Q, Sejling AS, Tiniakos D, Harrison SA. Artificial intelligence scoring of liver biopsies in a phase II trial of semaglutide in nonalcoholic steatohepatitis. Hepatology. 2024 Jul 1;80(1):173-185. doi: 10.1097/HEP.0000000000000723. Epub 2023 Dec 19. PMID 38112484
- [Derived] Wai-Sun Wong V, Anstee QM, Nitze LM, Geerts A, George J, Nolasco V, Kjaer MS, Ladelund S, Newsome PN, Ratziu V. FibroScan-aspartate aminotransferase (FAST) score for monitoring histological improvement in non-alcoholic steatohepatitis activity during semaglutide treatment: post-hoc analysis of a randomised, double-blind, placebo-controlled, phase 2b trial. EClinicalMedicine. 2023 Nov 20;66:102310. doi: 10.1016/j.eclinm.2023.102310. eCollection 2023 Dec. PMID 38058795
- [Derived] Romero-Gomez M, Armstrong MJ, Funuyet-Salas J, Mangla KK, Ladelund S, Sejling AS, Shrestha I, Sanyal AJ. Improved health-related quality of life with semaglutide in people with non-alcoholic steatohepatitis: A randomised trial. Aliment Pharmacol Ther. 2023 Aug;58(4):395-403. doi: 10.1111/apt.17598. Epub 2023 Jun 16. PMID 37328931
- [Derived] Harrison SA, Calanna S, Cusi K, Linder M, Okanoue T, Ratziu V, Sanyal A, Sejling AS, Newsome PN. Semaglutide for the treatment of non-alcoholic steatohepatitis: Trial design and comparison of non-invasive biomarkers. Contemp Clin Trials. 2020 Oct;97:106174. doi: 10.1016/j.cct.2020.106174. Epub 2020 Oct 8. PMID 33039693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 114 sites in 16 countries as follows (number of sites that screened participants/ number of sites that randomised participants): Australia (4/ 3); Austria (3/ 3); Belgium (4/ 4); Bulgaria (2/ 2); Canada (9/ 7); Denmark (2/ 2); Finland (1/ 1); France (8/ 6); Greece (5/ 5); Japan (13/ 12); Netherlands (7/ 5); Russian Federation (25/ 17); Spain (6/ 5); Sweden (3/ 2); United Kingdom (15/ 11); United States (36/ 29).
Pre-assignment Details: Participants were randomised in a 3:3:3:1:1:1 ratio to receive once-daily semaglutide or placebo subcutaneously. After randomisation, the participants entered a dose-escalation period, with increase in dose every 4 weeks until the target dose was reached.
Groups:
- Semaglutide 0.1 mg: Participants were to receive once daily subcutaneous (s.c.) injection of semaglutide for 72 weeks. Participants initially received 0.05 milligrams (mg) of semaglutide and the dose was then escalated once in 4 weeks until the target dose of 0.1 mg was reached: 0.05 mg (week 1 to week 4) and 0.1 mg (week 5 to week 72).
- Semaglutide 0.2 mg: Participants were to receive once daily s.c. injection of semaglutide for 72 weeks. Participants initially received 0.05 mg of semaglutide and the dose was then escalated once in 4 weeks until the target dose of 0.2 mg was reached: 0.05 mg (week 1 to week 4), 0.1 mg (week 5 to week 8) and 0.2 mg (week 9 to week 72).
- Semaglutide 0.4 mg: Participants were to receive once daily s.c. injection of semaglutide for 72 weeks. Participants initially received 0.05 mg of semaglutide and the dose was then escalated once in 4 weeks until the target dose of 0.4 mg was reached: 0.05 mg (week 1 to week 4), 0.1 mg (week 5 to week 8), 0.2 mg (week 9 to week 12), 0.3 mg (week 13 to week 16) and 0.4 mg (week 17 to week 72).
- Placebo: Participants were to receive once daily s.c. injection of placebo matched to semaglutide (0.05 mg, 0.1 mg, 0.2 mg, 0.3 mg or 0.4 mg) for 72 weeks.
Period: Overall Study
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Started | 80 | 78 | 82 | 80
Full Analysis Set | 80 | 78 | 82 | 80
Safety Analysis Set | 80 | 78 | 81 | 80
Exposed | 80 | 78 | 81 | 80
Completed | 76 | 72 | 77 | 77
Not Completed | 4 | 6 | 5 | 3
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo | Total
Number analyzed (Participants) | 80 | 78 | 82 | 80 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.9) | 58.1 (9.9) | 54.3 (10.2) | 52.4 (10.8) | 55.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 47 | 44 | 194
  Male | 29 | 26 | 35 | 36 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 14 | 9 | 40
  Not Hispanic or Latino | 69 | 63 | 65 | 66 | 263
  Unknown or Not Reported | 4 | 5 | 3 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 0 | 3
  Asian | 10 | 12 | 14 | 12 | 48
  Black or African American | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 65 | 59 | 62 | 62 | 248
  Other | 0 | 0 | 1 | 1 | 2
  Not applicable | 4 | 5 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non- Alcoholic Steatohepatitis (NASH) Resolution Without Worsening of Fibrosis After 72 Weeks (Yes/No)
Description: NASH resolution defined by NASH clinical research network as lobular inflammation of 0 or 1 and hepatocellular ballooning reduced to 0; both criteria were necessary conditions. Hepatocellular ballooning ranges from 0-2; lobular inflammation ranges from 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation. Worsening of fibrosis defined by an increase in fibrosis at least one stage of Kleiner fibrosis classification: fibrosis stages range from 0-4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis). Endpoint was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: After 72 weeks
Population: Full analysis set included all randomised participants. Overall number of participants analysed = Number of participants with fibrosis stage 2 or 3 at baseline who contributed to the analysis. In below table, 'Yes' infers percentage of participants who achieved NASH resolution without worsening of fibrosis and 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 57 | 59 | 56 | 58
Percentage of participants
  Yes | 40.4 | 35.6 | 58.9 | 17.2
  No | 54.4 | 47.5 | 30.4 | 74.1
  Missing | 5.3 | 16.9 | 10.7 | 8.6

2. Secondary Outcome: Percentage of Participants With at Least One Stage of Liver Fibrosis Improvement With no Worsening of NASH After 72 Weeks (Yes/No)
Description: NASH resolution defined by NASH clinical research network as lobular inflammation of 0 or 1; hepatocellular ballooning reduced to 0; both criteria were necessary conditions. Hepatocellular ballooning range: 0-2; lobular inflammation range: 0-3, with higher scores indicating more severe hepatocellular ballooning or lobular inflammation. Worsening of fibrosis defined by an increase in fibrosis at least one stage of Kleiner fibrosis classification: fibrosis stages range from 0-4, higher scores indicate greater fibrosis (0=None, 4=Cirrhosis). Endpoint was evaluated based on data from in-trial period which started on date of randomisation visit and ended on first of following dates (both inclusive):1) follow-up visit (Week 79); 2) withdrawal of consent; 3)last contact with participant (for participants lost to follow-up); 4)death.
Time Frame: After 72 weeks
Population: Full analysis set included all randomised participants. Overall number of participants analysed = Number of participants with fibrosis stage 2 or 3 at baseline who contributed to the analysis. In below table, 'Yes' infers percentage of participants who achieved at least one stage of fibrosis improvement with no worsening of NASH; 'No' infers vice-versa; 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 57 | 59 | 56 | 58
Percentage of participants
  Yes | 49.1 | 32.2 | 42.9 | 32.8
  No | 45.6 | 50.8 | 46.4 | 58.6
  Missing | 5.3 | 16.9 | 10.7 | 8.6

3. Secondary Outcome: Percentage of Participants With Change in Total NAFLD (Non- Alcoholic Fatty Liver Disease) Activity Score (NAS)
Description: Percentage of participants who had worsened, improved or had no change in total NAS from baseline to week 72 is presented. Worsening is defined as an increase of at least 1 in the NAS; Improvement is defined as a decrease of at least 1 in the NAS; while no change corresponds to no change in NAS from baseline to week 72. NAS is calculated as the sum of scores for steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocyte ballooning (0 to 2). Therefore, it is assessed on a scale of 0-8, with higher scores indicating more severe disease. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 71.3 | 79.5 | 82.9 | 43.8
  Worsening | 7.5 | 2.6 | 3.7 | 16.3
  No change | 13.8 | 5.1 | 1.2 | 27.5
  Missing | 7.5 | 12.8 | 12.2 | 12.5

4. Secondary Outcome: Percentage of Participants With Change in Steatosis
Description: Percentage of participants who had improved, worsened, or had no change in steatosis from baseline to week 72 is presented. Steatosis was assessed on a scale of 0-3, with higher scores indicating more severe steatosis. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 52.5 | 60.3 | 63.4 | 26.3
  Worsening | 6.3 | 2.6 | 3.7 | 15.0
  No change | 33.8 | 24.4 | 20.7 | 46.3
  Missing | 7.5 | 12.8 | 12.2 | 12.5

5. Secondary Outcome: Percentage of Participants With Change in Lobular Inflammation
Description: Percentage of participants who had improved, worsened, or had no change in lobular inflammation from baseline to week 72 is presented. Lobular inflammation was assessed on a scale of 0-3, with higher scores indicating more severe lobular inflammation. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 41.3 | 47.4 | 37.8 | 26.3
  Worsening | 7.5 | 7.7 | 6.1 | 17.5
  No change | 43.8 | 32.1 | 43.9 | 45.0
  Missing | 7.5 | 12.8 | 12.2 | 11.3

6. Secondary Outcome: Percentage of Participants With Change in Hepatocyte Ballooning
Description: Percentage of participants who had improved, worsened, or had no change in hepatocyte ballooning from baseline to week 72 is presented. Hepatocyte ballooning was assessed on a scale of 0-2, with higher scores indicating more severe disease. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 61.3 | 70.5 | 74.4 | 38.8
  Worsening | 2.5 | 2.6 | 1.2 | 2.5
  No change | 28.8 | 14.1 | 12.2 | 46.3
  Missing | 7.5 | 12.8 | 12.2 | 12.5

7. Secondary Outcome: Percentage of Participants With Change in Fibrosis Stage According to the Kleiner Fibrosis Classification
Description: Percentage of participants who had improved, worsened, or had no change in fibrosis stage from baseline to week 72 is presented. The degree of fibrosis is described by the Kleiner fibrosis staging system, ranging from F0 (absence of fibrosis), F1 (portal/perisinusoidal fibrosis), F2 (perisinusoidal and portal/periportal fibrosis), F3 (septal or bridging fibrosis) through F4 (cirrhosis). The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 46.3 | 32.1 | 42.7 | 31.3
  Worsening | 10.0 | 7.7 | 4.9 | 18.8
  No change | 36.3 | 42.3 | 36.6 | 37.5
  Missing | 7.5 | 17.9 | 15.9 | 12.5

8. Secondary Outcome: Percentage of Participants With Change in Activity Component of Steatosis-activity-fibrosis (SAF) Score
Description: Percentage of participants who had improved, worsened, or had no change in the activity component of the SAF score from baseline to week 72 is presented. SAF score was assessed on a scale of 0-4, with higher scores indicating more severe disease. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Improvement | 62.5 | 71.8 | 72.0 | 42.5
  Worsening | 7.5 | 3.8 | 1.2 | 11.3
  No change | 22.5 | 11.5 | 14.6 | 33.8
  Missing | 7.5 | 12.8 | 12.2 | 12.5

9. Secondary Outcome: Change in Fibrosis-4 Score
Description: Change in fibrosis-4 score is presented as ratio to baseline. Fibrosis-4 is the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, alanine aminotransferase (ALT), AST and age that is calculated using formula: Fibrosis-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A Fibrosis-4 index of < 1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants. Overall number of participants analysed = Number of participants who contributed to the analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fibrosis-4 score
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 63 | 72 | 67
Ratio of fibrosis-4 score | 0.81 (36.8) | 0.77 (32.4) | 0.77 (31.3) | 0.95 (43.1)

10. Secondary Outcome: Change in NAFLD Fibrosis Score (NFS)
Description: Change in NFS from baseline to week 72 is presented. NFS is calculated using formula: NFS = -1.675 + 0.037 * age (years) + 0.094 * body mass index (BMI) (kg/m^2) + 1.13 * hyperglycaemia (yes/no) + 0.99 * Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) ratio + 0.013 × platelet count (*10^9/L) - 0.66 * albumin (g/dL). The score is used to classify the probability of fibrosis. A score a) < -1.5 indicates a low probability, b) > -1.5 to < 0.67 indicates intermediate probability, and a score of c) > 0.67 indicates a high probability of liver fibrosis. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 63 | 72 | 66
Score on a scale | -0.322 (0.819) | -0.617 (0.691) | -0.475 (0.770) | -0.040 (0.844)

11. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Change in ALT (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALT
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 75
Ratio of ALT | 0.62 (62.7) | 0.57 (62.1) | 0.40 (68.2) | 0.80 (60.3)

12. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Change in AST (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AST
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 69 | 77 | 74
Ratio of AST | 0.66 (55.1) | 0.63 (46.6) | 0.50 (45.8) | 0.84 (62.3)

13. Secondary Outcome: Change in Gamma Glutamyl Transferase (GGT)
Description: Change in GGT (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of GGT
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 75
Ratio of GGT | 0.76 (52.0) | 0.64 (51.6) | 0.48 (60.2) | 0.92 (46.6)

14. Secondary Outcome: Change in Albumin
Description: Change in albumin (measured as grams per deciliter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 75
Ratio of albumin | 1.02 (5.6) | 1.01 (6.0) | 1.01 (5.4) | 1.02 (6.0)

15. Secondary Outcome: Change in International Normalized Ratio (INR)
Description: Change in INR is presented as ratio to baseline. INR is the ratio of measured prothrombin time over normal prothrombin time and it evaluates the extrinsic coagulation pathway (vitamin K dependent clotting factors II; V, VII, IX and X). These clotting factors are synthesised in the liver, thus INR is used as a marker of liver synthesis function. The therapeutic INR range varies, most commonly an INR 2-3 goal, but ranging from 1.5-4.0. Bleeding complications are more likely to occur above an INR value of 4.0. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of INR
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 76 | 75
Ratio of INR | 0.97 (18.8) | 0.96 (11.8) | 0.93 (22.3) | 0.99 (19.3)

16. Secondary Outcome: Change in Enhanced Liver Fibrosis (ELF)
Description: Change in ELF from baseline to week 72 is presented. The ELF discriminant score was derived as a log-linear combination of the markers hyaluronic acid (HA), amino-terminal propeptide of type III collagen (PIIINP) and tissue inhibitor of metalloproteinase 1 (TIMP1). ELF score = -7.412 + 0.681 × ln(HA (nanograms per millilitre (ng/mL)) + 0.775 × ln(P3NP (ng/mL)) + 0.494 × ln(TIMP1 (ng/mL)). ELF score: a) < 7.7: no to mild fibrosis; b) ≥ 7.7 - < 9.8: Moderate fibrosis; c) ≥ 9.8 - < 11.3: Severe fibrosis; d) ≥ 11.3: Cirrhosis. A negative change from baseline indicates decreased fibrosis. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 70 | 76 | 75
score on a scale | -0.4 (0.7) | -0.4 (0.8) | -0.6 (0.8) | 0.1 (0.7)

17. Secondary Outcome: Change in Cytokeratin 18 (CK-18) Fragments
Description: Change in CK-18 fragments (M30, M65) (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of CK-18 fragments
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 76 | 74
Ratio of CK-18 fragments
  M30 | 0.52 (84.2) | 0.50 (76.4) | 0.40 (74.5) | 0.78 (106.9)
  M65 | 0.51 (73.1) | 0.52 (62.5) | 0.38 (65.6) | 0.71 (83.7)

18. Secondary Outcome: Change in microRNA 122 (miR-122)
Description: Change in miR-122 (measured as 1/microliter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.Overall number of participants analysed = Number of participants who contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of miR-122
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 73 | 71 | 76 | 74
Ratio of miR-122 | 0.86 (151.8) | 0.74 (203.1) | 0.58 (161.3) | 1.28 (194.3)

19. Secondary Outcome: Change in Interleukin-1 Receptor (IL-1R) Antagonist
Description: Change in interleukin-1 receptor (IL-1R) antagonist (measured as picograms per milliliter) antagonist is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of IL-1R antagonist
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 69 | 65 | 74 | 69
Ratio of IL-1R antagonist | 0.87 (49.3) | 0.85 (37.5) | 0.73 (47.9) | 0.94 (41.7)

20. Secondary Outcome: Change in Monocyte Chemoattractant Protein 1 (MCP-1)
Description: Change in MCP-1 (measured as picograms per milliliter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of MCP-1
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 75 | 71 | 76 | 73
Ratio of MCP-1 | 1.07 (23.3) | 1.08 (29.8) | 0.99 (30.7) | 1.04 (26.4)

21. Secondary Outcome: Change in Fibroblast Growth Factor 21 (FGF-21)
Description: Change in FGF-21 (measured as picograms per milliliter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FGF-21
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 74
Ratio of FGF-21 | 0.72 (86.1) | 0.61 (104.1) | 0.55 (91.3) | 0.76 (64.8)

22. Secondary Outcome: Change in Liver Stiffness Assessed by FibroScan®
Description: Change in liver stiffness (measured as kilopascal (kPa)) assessed by FibroScan® is presented as ratio to baseline. FibroScan® is a specialized ultrasound machine for the liver. It measures fibrosis (scarring) by measuring the stiffness of the liver. It's normally between 2 and 6 kPa. Many people with liver disease(s) have a result that's higher than the normal range. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of liver stiffness
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 47 | 49 | 46 | 45
Ratio of liver stiffness | 0.72 (49.3) | 0.64 (52.2) | 0.66 (58.4) | 1.18 (71.2)

23. Secondary Outcome: Change in Liver Steatosis Assessed by FibroScan®
Description: Change in liver steatosis assessed by FibroScan® from baseline to week 72 is presented. FibroScan® is a specialized ultrasound machine for the liver. It measures fibrosis (scarring) and steatosis (fatty change) in the liver. Fatty change is fat building up in the liver cells. To assess liver steatosis, the controlled attenuation parameter (CAP; giving an estimate of ultrasound attenuation ∼3.5 MegaHertz (MHz)) is available with the M probe of the FibroScan. The CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m, with higher scores indicating higher amount of liver with fatty change. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Decibels per meter
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 34 | 37 | 33 | 35
Decibels per meter | -5.8 (41.1) | -50.9 (64.3) | -42.1 (73.3) | -18.7 (43.3)

24. Secondary Outcome: Percentage of Participants With Weight Loss of ≥ 5% of Baseline Body Weight at 72 Weeks (Yes/No)
Description: Percentage of participants with weight loss of greater than or equal to (≥) 5% of baseline body weight at 72 weeks is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death. In the below table, 'Yes' infers percentage of participants who have achieved ≥ 5% weight loss; 'No' infers percentage of participants who have not achieved ≥ 5% weight loss at 72 weeks and 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Time Frame: Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Yes | 43.8 | 62.8 | 76.8 | 16.3
  No | 51.3 | 28.2 | 17.1 | 78.8
  Missing | 5.0 | 9.0 | 6.1 | 5.0

25. Secondary Outcome: Percentage of Participants With Weight Loss of ≥ 10% of Baseline Body Weight at 72 Weeks (Yes/No)
Description: Pentage of participants with weight loss of ≥ 10% of baseline body weight at 72 weeks is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death. In the below table, 'Yes' infers percentage of participants who have achieved ≥ 10% weight loss; 'No' infers percentage of participants who have not achieved ≥ 10% weight loss at 72 weeks and 'Missing' refers to percentage of participants with data missing due to different reasons (lost to follow-up, withdrawal).
Time Frame: Week 72
Population: Full analysis set included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Percentage of participants
  Yes | 17.5 | 38.5 | 59.8 | 2.5
  No | 77.5 | 52.6 | 34.1 | 92.5
  Missing | 5.0 | 9.0 | 6.1 | 5.0

26. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 76
Kilograms | -4.8 (6.0) | -9.4 (9.2) | -12.3 (8.6) | -1.0 (4.9)

27. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 69 | 77 | 75
Centimeters | -3.9 (6.3) | -7.1 (8.9) | -11.4 (9.3) | -1.7 (6.2)

28. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Kilograms per square meter
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 76
Kilograms per square meter | -1.8 (2.2) | -3.5 (3.4) | -4.6 (3.3) | -0.3 (1.8)

29. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) (%-Point)
Description: Change in HbA1c (measured as percentage point of HbA1c) from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants. Overall number of participants analysed = Number of participants with type 2 diabetes who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 47
Percentage point of HbA1c | -0.7 (1.1) | -1.2 (0.9) | -1.2 (1.0) | -0.0 (1.0)

30. Secondary Outcome: Change in HbA1c (Millimoles Per Mole)
Description: Change in HbA1c from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: millimoles per mole
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 46 | 45 | 47 | 47
millimoles per mole | -7.9 (12.2) | -12.8 (9.5) | -12.8 (11.3) | -0.3 (10.7)

31. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 47 | 48
Millimoles per liter | -1.39 (2.53) | -2.17 (1.82) | -2.09 (2.68) | -0.34 (2.72)

32. Secondary Outcome: Change in Fasting Glucagon
Description: Change in fasting glucagon (measured as picograms per milliliter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of glucagon
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 45 | 45 | 47 | 47
Ratio of glucagon | 0.78 (76.8) | 0.65 (94.8) | 0.63 (100.4) | 1.04 (80.8)

33. Secondary Outcome: Change in Homeostatic Model Assessment - Insulin Resistance (HOMA-IR)
Description: Change in HOMA-IR is presented as ratio to baseline. HOMA-IR was calculated as: Insulin resistance (%) = fasting plasma glucose [mmol/L] x fasting insulin [mmol/L]/ 22.5. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: Full analysis set included all randomised participants.Overall number of participants analysed = Number of participants with type 2 diabetes who contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-IR
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 42 | 43 | 44 | 45
Ratio of HOMA-IR | 0.77 (62.2) | 0.60 (77.6) | 0.58 (94.6) | 0.81 (127.5)

34. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in a sitting position after 5 minutes of rest. Change in DBP from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 70 | 77 | 76
Millimeters of mercury | 0 (10) | -2 (11) | -2 (9) | -1 (10)

35. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Blood pressure was measured in a sitting position after 5 minutes of rest. Change in SBP from baseline to week 72 is presented. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 70 | 77 | 76
Millimeters of mercury | -2 (16) | -7 (18) | -6 (16) | -2 (15)

36. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 75 | 68 | 77 | 75
Ratio of total cholesterol | 0.98 (17.1) | 1.00 (20.3) | 0.93 (15.7) | 0.93 (18.8)

37. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Change in LDL cholesterol (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 73 | 68 | 77 | 75
Ratio of LDL cholesterol | 0.96 (22.9) | 1.01 (34.9) | 0.92 (25.5) | 0.90 (30.7)

38. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol
Description: Change in HDL cholesterol (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 68 | 77 | 75
Ratio of HDL cholesterol | 1.04 (16.1) | 1.05 (12.9) | 1.09 (16.4) | 1.01 (12.9)

39. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL) Cholesterol
Description: Change in VLDL cholesterol (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 73 | 68 | 77 | 75
Ratio of VLDL cholesterol | 0.89 (31.9) | 0.90 (36.1) | 0.74 (38.2) | 0.93 (36.7)

40. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 68 | 77 | 75
Ratio of triglycerides | 0.88 (34.1) | 0.89 (37.6) | 0.73 (41.4) | 0.95 (36.9)

41. Secondary Outcome: Change in Free Fatty Acids
Description: Change in free fatty acids (measured as millimoles per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 72 | 68 | 74 | 72
Ratio of free fatty acids | 0.83 (54.8) | 0.92 (73.2) | 0.72 (80.8) | 1.05 (75.9)

42. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)
Description: Change in hsCRP (measured as milligram per liter) from baseline to week 72 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 76 | 71 | 77 | 75
Ratio of hsCRP | 0.78 (114.6) | 0.50 (124.1) | 0.41 (114.6) | 0.91 (85.8)

43. Secondary Outcome: Change in Short Form 36 (SF-36) Score
Description: Change in SF-36 score from baseline to week 72 is presented. SF-36 measures participant's overall health related quality of life (HRQoL). It is a 36-item generic measure of health status and yields 2 summary scores for physical health and mental health, and 8 domain scores (physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional, mental health). The scores 0-100 (where higher scores indicates a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of scores in the 2009 U.S. general population. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 82 | 80
Scores on a scale
  Mental component sum: number analyzed (Participants) | 76 | 68 | 77 | 74
  Mental component sum | 2.2 (8.5) | 0.6 (9.2) | 1.2 (9.5) | -0.4 (8.9)
  Physical component sum: number analyzed (Participants) | 76 | 68 | 76 | 74
  Physical component sum | 2.1 (7.0) | 1.1 (7.3) | 3.9 (7.1) | -0.1 (8.3)
  Physical functioning: number analyzed (Participants) | 76 | 70 | 76 | 75
  Physical functioning | 1.8 (7.8) | 2.0 (7.3) | 2.8 (7.8) | -0.4 (8.2)
  Role functioning: number analyzed (Participants) | 76 | 69 | 77 | 74
  Role functioning | 2.1 (6.9) | 0.5 (9.3) | 2.2 (8.1) | -0.3 (9.4)
  Bodily pain: number analyzed (Participants) | 76 | 70 | 77 | 75
  Bodily pain | 1.3 (10.9) | 1.2 (10.1) | 3.4 (7.9) | -1.3 (10.2)
  General health: number analyzed (Participants) | 76 | 70 | 77 | 75
  General health | 7.2 (14.8) | 2.3 (17.8) | 9.0 (17.4) | 4.3 (16.5)
  Vitality: number analyzed (Participants) | 76 | 69 | 77 | 75
  Vitality | 2.3 (8.6) | 0.6 (9.4) | 4.6 (9.8) | -0.2 (10.1)
  Social functioning: number analyzed (Participants) | 76 | 70 | 77 | 75
  Social functioning | 3.7 (9.0) | -0.1 (9.9) | 2.2 (9.4) | -1.6 (8.3)
  Role emotional: number analyzed (Participants) | 76 | 68 | 77 | 74
  Role emotional | 2.2 (8.9) | 0.6 (9.1) | 0.5 (9.5) | -0.3 (8.5)
  Mental health: number analyzed (Participants) | 76 | 69 | 77 | 75
  Mental health | 1.2 (8.9) | 1.5 (8.2) | 1.3 (9.5) | -0.2 (9.7)

44. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant administered or using a medicinal product, whether or not considered related to the medicinal product or usage. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half lives of semaglutide); 2) end of the in-trial period.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Number; unit: events
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
events | 525 | 577 | 511 | 445

45. Secondary Outcome: Number of Treatment-emergent Hypoglycaemic Episodes
Description: Hypoglycaemic episode (blood glucose less than or equal to (<=) 3.9 mmol/L (70 mg/dL) Or greater than (>) 3.9 mmol/L (70 mg/dL) occurring in conjunction with hypoglycaemic symptoms) is defined as treatment emergent if the onset of the episode occurs during the on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment. Overall number of participants analysed = Number of participants with type 2 diabetes who contributed to the analysis.
Measure: Number; unit: episodes
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 49 | 50
episodes | 54 | 30 | 66 | 18

46. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose (BG)-Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemia: episode, severe as per american diabetes association (ADA) classification or BG confirmed by plasma glucose value < 3.1 mmol/L(56mg/dL) with symptoms along with hypoglycaemia. Severe hypoglycaemia: episode requiring assistance of other person to actively administer carbohydrate, glucagon, or take corrective actions. Plasma glucose concentrations may not be available during event, but neurological recovery following return of plasma glucose to normal is sufficient evidence that event was induced by low plasma glucose concentration. Hypoglycaemic episode is treatment emergent if onset of it occurs during on-treatment period: period starting on day of first administration of trial product and ending on day of last dose of trial product+7 days; except for evaluation of AEs; hypoglycaemic episodes for which period ended on date of whatever came first:last dose of trial product + 49 days (7 half-lives of semaglutide); end of in-trial period.
Time Frame: From week 0 to week 79
Population: as for outcome 45
Measure: Number; unit: episodes
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 49 | 50
episodes | 3 | 5 | 17 | 2

47. Secondary Outcome: Number of Treatment-emergent Severe Hypoglycaemic Episodes
Description: Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration. Hypoglycaemic episode is defined as treatment emergent if the onset of the episode occurs during the on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: From week 0 to week 79
Population: as for outcome 45
Measure: Number; unit: episodes
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 49 | 51 | 49 | 50
episodes | 2 | 2 | 0 | 0

48. Secondary Outcome: Number of Participants Discontinuing Treatment Due to Gastrointestinal Adverse Events
Description: Number of participants discontinuing treatment due to gastrointestinal adverse events is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Participants | 1 | 6 | 2 | 0

49. Secondary Outcome: Number of Participants With Occurrence of Anti-semaglutide Antibodies During and After 72 Weeks Treatment (Yes/No)
Description: Number of participants with occurrence of anti-semaglutide antibodies during and after 72 weeks treatment is presented. In the below table, 'Yes' infers number of participants with occurrence of anti-semaglutide antibodies and 'No' infers number of participants without anti-semaglutide antibodies during and after 72 weeks treatment. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg
Number analyzed (Participants) | 80 | 78 | 81
Participants
  Yes | 4 | 1 | 2
  No | 76 | 77 | 79

50. Secondary Outcome: Number of Participants With Anti-semaglutide Antibodies With in Vitro Neutralising Effect During and After 72 Weeks Treatment (Yes/No)
Description: Number of participants with anti-semaglutide antibodies with in vitro neutralising effect during and after 72 weeks treatment is presented. In the below table, 'Yes' infers number of participants with anti-semaglutide antibodies with in vitro neutralising effect and 'No' infers number of participants without anti-semaglutide antibodies with in vitro neutralising effect during and after 72 weeks treatment. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg
Number analyzed (Participants) | 80 | 78 | 81
Participants
  Yes | 0 | 0 | 0
  No | 80 | 78 | 81

51. Secondary Outcome: Number of Participants With Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 During and After 72 Weeks Treatment (Yes/No)
Description: Number of participants with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) during and after 72 weeks treatment is presented. In the below table, 'Yes' infers number of participants with anti-semaglutide antibodies cross reacting with native GLP-1 and 'No' infers number of participants without anti-semaglutide antibodies cross reacting with native GLP-1 during and after 72 weeks treatment. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg
Number analyzed (Participants) | 80 | 78 | 81
Participants
  Yes | 4 | 0 | 2
  No | 76 | 78 | 79

52. Secondary Outcome: Number of Participants With Cross-reacting Anti-semaglutide Binding Antibodies With in Vitro Neutralising Effect to Native GLP-1 During and After 72 Weeks Treatment (Yes/No)
Description: Number of participants with cross-reacting anti-semaglutide binding antibodies with in vitro neutralising effect to native GLP-1 during and after 72 weeks treatment is presented. In the below table, 'Yes' infers number of participants with cross-reacting anti-semaglutide binding antibodies with in vitro neutralising effect to native GLP-1 and 'No' infers number of participants without cross-reacting anti-semaglutide binding antibodies with in vitro neutralising effect to native GLP-1 during and after 72 weeks treatment. The endpoint was evaluated based on the data from in-trial period which started on the date of the randomisation visit and ended on the first of the following dates (both inclusive): 1) follow-up visit (Week 79); 2) withdrawal of consent; 3) last contact with participant (for participants lost to follow-up); 4) death.
Time Frame: From week 0 to week 79
Population: Safety analysis set included all participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg
Number analyzed (Participants) | 80 | 78 | 81
Participants
  Yes | 0 | 0 | 0
  No | 80 | 78 | 81

53. Secondary Outcome: Change in Pulse From Baseline to Week 72
Description: Change in pulse from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: Safety analysis set included all participants who received at least one dose of randomised treatment. Overall number of participants analysed = Number of participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 73 | 63 | 72 | 71
beats per minute (bpm) | 2.2 (10.9) | 2.1 (9.0) | 0.9 (9.6) | -0.3 (9.1)

54. Secondary Outcome: Percentage of Participants With Change in Electrocardiogram (ECG)
Description: A 12-lead ECG was performed at baseline (week 0) and week 72 and categorised as normal, abnormal and not clinically significant (abnormal NCS) or abnormal and clinically significant (abnormal CS). Percentage of participants in each ECG category at week 0 and week 72 are presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Percentage of participants
  Week 0: Normal | 58.8 | 60.3 | 66.7 | 63.8
  Week 0: Abnormal NCS | 41.3 | 39.7 | 32.1 | 36.3
  Week 0: Abnormal CS | 0.0 | 0.0 | 1.2 | 0.0
  Week 72: Normal: number analyzed (Participants) | 74 | 63 | 71 | 70
  Week 72: Normal | 64.9 | 65.1 | 74.6 | 60.0
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 63 | 71 | 70
  Week 72: Abnormal NCS | 35.1 | 34.9 | 23.9 | 38.6
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 63 | 71 | 70
  Week 72: Abnormal CS | 0.0 | 0.0 | 1.4 | 1.4

55. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Cardiovascular System
Description: Percentage of participants with change in physical examination (cardiovascular system) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Percentage of participants
  Week -6: Normal | 87.5 | 93.6 | 92.6 | 92.5
  Week -6: Abnormal NCS | 11.3 | 5.1 | 7.4 | 6.3
  Week -6: Abnormal CS | 1.3 | 1.3 | 0.0 | 1.3
  Week 72: Normal: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Normal | 87.8 | 96.9 | 94.4 | 90.1
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal NCS | 12.2 | 3.1 | 5.6 | 8.5
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal CS | 0.0 | 0.0 | 0.0 | 1.4

56. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Central and Peripheral Nervous System
Description: Percentage of participants with change in physical examination (central and peripheral nervous system) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 79 | 80
Percentage of participants
  Week -6: Normal | 92.5 | 94.8 | 98.7 | 95.0
  Week -6: Abnormal NCS | 5.0 | 5.2 | 1.3 | 3.8
  Week -6: Abnormal CS | 2.5 | 0.0 | 0.0 | 1.3
  Week 72: Normal: number analyzed (Participants) | 74 | 63 | 69 | 70
  Week 72: Normal | 94.6 | 93.7 | 98.6 | 92.9
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 63 | 69 | 70
  Week 72: Abnormal NCS | 5.4 | 4.8 | 1.4 | 7.1
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 63 | 69 | 70
  Week 72: Abnormal CS | 0.0 | 1.6 | 0.0 | 0.0

57. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Gastrointestinal System Including Mouth
Description: Percentage of participants with change in physical examination (gastrointestinal system including mouth) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 81 | 80
Percentage of participants
  Week -6: Normal | 82.5 | 83.1 | 84.0 | 86.3
  Week -6: Abnormal NCS | 13.8 | 15.6 | 16.0 | 12.5
  Week -6: Abnormal CS | 3.8 | 1.3 | 0.0 | 1.3
  Week 72: Normal: number analyzed (Participants) | 74 | 63 | 72 | 71
  Week 72: Normal | 89.2 | 81.0 | 87.5 | 84.5
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 63 | 72 | 71
  Week 72: Abnormal NCS | 10.8 | 19.0 | 12.5 | 14.1
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 63 | 72 | 71
  Week 72: Abnormal CS | 0.0 | 0.0 | 0.0 | 1.4

58. Secondary Outcome: Percentage of Participants With Change in Physical Examination: General Appearance
Description: Percentage of participants with change in physical examination (general appearance) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Percentage of participants
  Week -6: Normal | 83.8 | 85.9 | 79.0 | 80.0
  Week -6: Abnormal NCS | 16.3 | 12.8 | 21.0 | 20.0
  Week -6: Abnormal CS | 0.0 | 1.3 | 0.0 | 0.0
  Week 72: Normal: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Normal | 83.8 | 90.6 | 90.3 | 76.1
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal NCS | 16.2 | 6.3 | 9.7 | 23.9
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal CS | 0.0 | 3.1 | 0.0 | 0.0

59. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Head, Ears, Eyes, Nose, Throat, Neck
Description: Percentage of participants with change in physical examination (head, ears, eyes, nose, throat, neck) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 80 | 80
Percentage of participants
  Week -6: Normal | 97.5 | 94.8 | 98.8 | 97.5
  Week -6: Abnormal NCS | 2.5 | 5.2 | 1.3 | 2.5
  Week -6: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: Normal: number analyzed (Participants) | 73 | 62 | 70 | 71
  Week 72: Normal | 94.5 | 96.8 | 98.6 | 98.6
  Week 72: Abnormal NCS: number analyzed (Participants) | 73 | 62 | 70 | 71
  Week 72: Abnormal NCS | 4.1 | 3.2 | 1.4 | 0.0
  Week 72: Abnormal CS: number analyzed (Participants) | 73 | 62 | 70 | 71
  Week 72: Abnormal CS | 1.4 | 0.0 | 0.0 | 1.4

60. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Lymph Node Palpation
Description: Percentage of participants with change in physical examination (lymph node palpation) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 78 | 80
Percentage of participants
  Week -6: Normal | 100.0 | 98.7 | 100.0 | 100.0
  Week -6: Abnormal NCS | 0.0 | 1.3 | 0.0 | 0.0
  Week -6: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: Normal: number analyzed (Participants) | 74 | 60 | 70 | 71
  Week 72: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 60 | 70 | 71
  Week 72: Abnormal NCS | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 60 | 70 | 71
  Week 72: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0

61. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Musculoskeletal System
Description: Percentage of participants with change in physical examination (musculoskeletal system) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 79 | 80
Percentage of participants
  Week -6: Normal | 95.0 | 96.1 | 94.9 | 95.0
  Week -6: Abnormal NCS | 3.8 | 3.9 | 5.1 | 3.8
  Week -6: Abnormal CS | 1.3 | 0.0 | 0.0 | 1.3
  Week 72: Normal: number analyzed (Participants) | 74 | 63 | 70 | 71
  Week 72: Normal | 94.6 | 96.8 | 100.0 | 95.8
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 63 | 70 | 71
  Week 72: Abnormal NCS | 5.4 | 3.2 | 0.0 | 4.2
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 63 | 70 | 71
  Week 72: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0

62. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Respiratory System
Description: Percentage of participants with change in physical examination (respiratory system) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Percentage of participants
  Week -6: Normal | 100.0 | 100.0 | 100.0 | 97.5
  Week -6: Abnormal NCS | 0.0 | 0.0 | 0.0 | 2.5
  Week -6: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: Normal: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Normal | 98.6 | 96.9 | 98.6 | 98.6
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal NCS | 0.0 | 3.1 | 1.4 | 1.4
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 64 | 72 | 71
  Week 72: Abnormal CS | 1.4 | 0.0 | 0.0 | 0.0

63. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Skin
Description: Percentage of participants with change in physical examination (skin) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 78 | 81 | 80
Percentage of participants
  Week -6: Normal | 96.3 | 92.3 | 85.2 | 90.0
  Week -6: Abnormal NCS | 2.5 | 6.4 | 13.6 | 10.0
  Week -6: Abnormal CS | 1.3 | 1.3 | 1.2 | 0.0
  Week 72: Normal: number analyzed (Participants) | 74 | 64 | 70 | 71
  Week 72: Normal | 94.6 | 87.5 | 90.0 | 88.7
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 64 | 70 | 71
  Week 72: Abnormal NCS | 4.1 | 10.9 | 8.6 | 11.3
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 64 | 70 | 71
  Week 72: Abnormal CS | 1.4 | 1.6 | 1.4 | 0.0

64. Secondary Outcome: Percentage of Participants With Change in Physical Examination: Thyroid Gland
Description: Percentage of participants with change in physical examination (thyroid gland) from week -6 to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Week -6, week 72
Population: as for outcome 53
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 80 | 77 | 80 | 80
Percentage of participants
  Week -6: Normal | 88.8 | 97.4 | 97.5 | 98.8
  Week -6: Abnormal NCS | 10.0 | 2.6 | 2.5 | 0.0
  Week -6: Abnormal CS | 1.3 | 0.0 | 0.0 | 1.3
  Week 72: Normal: number analyzed (Participants) | 74 | 62 | 70 | 70
  Week 72: Normal | 94.6 | 98.4 | 97.1 | 98.6
  Week 72: Abnormal NCS: number analyzed (Participants) | 74 | 62 | 70 | 70
  Week 72: Abnormal NCS | 5.4 | 1.6 | 2.9 | 1.4
  Week 72: Abnormal CS: number analyzed (Participants) | 74 | 62 | 70 | 70
  Week 72: Abnormal CS | 0.0 | 0.0 | 0.0 | 0.0

65. Secondary Outcome: Change in Haematocrit
Description: Change in haematocrit from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Percentage of haematocrit in blood
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 70 | 68
Percentage of haematocrit in blood | -0.79 (3.14) | -0.71 (2.77) | -1.43 (3.50) | -0.41 (3.53)

66. Secondary Outcome: Change in Haemoglobin (g/dL)
Description: Change in haemoglobin from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 70 | 68
Grams per deciliter (g/dL) | 0.18 (1.05) | 0.08 (0.89) | -0.07 (0.98) | 0.21 (1.08)

67. Secondary Outcome: Change in Haemoglobin (mmol/L)
Description: as for outcome 66
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 70 | 68
millimoles per liter (mmol/L) | 0.11 (0.65) | 0.05 (0.55) | -0.05 (0.61) | 0.13 (0.67)

68. Secondary Outcome: Change in Leukocytes
Description: Change in leukocytes from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 70 | 68
10^9 cells per liter (10^9/L) | 0.489 (1.564) | 0.260 (1.343) | -0.047 (1.532) | 0.075 (1.733)

69. Secondary Outcome: Change in Thrombocytes
Description: Change in thrombocytes from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 69 | 67
10^9 cells per liter (10^9/L) | 8.8 (46.9) | 14.6 (34.8) | 9.0 (44.9) | 0.3 (43.7)

70. Secondary Outcome: Change in Erythrocytes
Description: Change in erythrocytes from baseline to week 72 is presented. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12/L)
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 71 | 59 | 70 | 68
10^12 cells per liter (10^12/L) | 0.038 (0.292) | 0.004 (0.220) | -0.034 (0.334) | 0.054 (0.314)

71. Secondary Outcome: Change in Creatinine (mg/dL)
Description: Change in creatinine (measured as milligram per deciliter (mg/dL)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatinine
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of creatinine | 1.018 (30.70) | 1.069 (42.19) | 1.026 (35.17) | 1.021 (33.87)

72. Secondary Outcome: Change in Creatinine (Umol/L)
Description: Change in creatinine (measured as micro mole per liter (umol/L)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatinine
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of creatinine | 1.018 (30.70) | 1.069 (42.19) | 1.026 (35.17) | 1.021 (33.87)

73. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change in eGFR (measured as milliliter/minute/1.732 meter square (mL/min/1.73 m^2)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of eGFR
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of eGFR | 0.976 (28.04) | 0.940 (40.47) | 0.973 (31.42) | 0.969 (31.24)

74. Secondary Outcome: Change in Creatine Kinase
Description: Change in creatine kinase (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of creatine kinase
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of creatine kinase | 0.975 (73.02) | 0.798 (77.96) | 0.825 (74.17) | 0.904 (76.04)

75. Secondary Outcome: Change in Urea
Description: Change in urea (measured as milli mole per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of urea
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of urea | 1.018 (51.01) | 0.973 (52.30) | 1.042 (51.14) | 1.043 (52.30)

76. Secondary Outcome: Change in Total Bilirubin (mg/dL)
Description: Change in total bilirubin (measured as milligram per deciliter (mg/dL)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of total bilirubin | 0.978 (66.72) | 1.011 (70.66) | 0.949 (65.89) | 1.040 (67.36)

77. Secondary Outcome: Change in Total Bilirubin (Umol/L)
Description: Change in total bilirubin (measured as micromole per liter (umol/L)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total bilirubin
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of total bilirubin | 0.978 (66.72) | 1.011 (70.66) | 0.949 (65.89) | 1.040 (67.36)

78. Secondary Outcome: Change in Alkaline Phosphatase
Description: Change in alkaline phosphatase (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of alkaline phosphatase
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of alkaline phosphatase | 0.980 (45.68) | 0.931 (43.59) | 0.884 (54.90) | 0.992 (42.42)

79. Secondary Outcome: Change in Ferritin
Description: Change in ferritin (measured as microgram per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ferritin
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of ferritin | 0.660 (99.95) | 0.617 (88.70) | 0.603 (88.83) | 0.713 (96.91)

80. Secondary Outcome: Change in Sodium (mEq/L)
Description: Change in sodium (measured as milli equivalent per liter (mEq/L)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of sodium | 0.999 (12.23) | 1.000 (12.13) | 1.002 (11.68) | 1.002 (12.91)

81. Secondary Outcome: Change in Sodium (mmol/L)
Description: Change in sodium (measured as milli mole per liter (mmol/L)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of sodium | 0.999 (12.23) | 1.000 (12.13) | 1.002 (11.68) | 1.002 (12.91)

82. Secondary Outcome: Change in Potassium (mEq/L)
Description: Change in potassium (measured as mEq/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 61 | 72 | 69
Ratio of potassium | 1.004 (27.00) | 0.979 (29.36) | 0.998 (27.81) | 0.998 (27.78)

83. Secondary Outcome: Change in Potassium (mmol/L)
Description: Change in potassium (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 61 | 72 | 69
Ratio of potassium | 1.004 (27.00) | 0.979 (29.36) | 0.998 (27.81) | 0.998 (27.78)

84. Secondary Outcome: Change in Calcium (mg/dL)
Description: Change in calcium (measured as milligram per deciliter (mg/dL)) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of calcium | 1.017 (20.37) | 1.018 (20.49) | 1.008 (20.88) | 1.010 (22.79)

85. Secondary Outcome: Change in Calcium (mmol/L)
Description: Change in calcium (measured as mmol/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of calcium | 1.017 (20.37) | 1.018 (20.49) | 1.008 (20.88) | 1.010 (22.79)

86. Secondary Outcome: Change in Amylase
Description: Change in amylase (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of amylase | 1.155 (49.85) | 1.120 (65.01) | 1.170 (47.88) | 1.051 (45.74)

87. Secondary Outcome: Change in Lipase
Description: Change in lipase (measured as units per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of lipase | 1.305 (77.43) | 1.245 (87.68) | 1.375 (73.88) | 1.003 (66.72)

88. Secondary Outcome: Change in Calcitonin
Description: Change in calcitonin (measured as nanograms per liter) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half-lives of semaglutide); 2) end of the in-trial period.
Time Frame: Baseline (week 0), Week 72
Population: as for outcome 53
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Calcitonin
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
Number analyzed (Participants) | 74 | 62 | 72 | 70
Ratio of Calcitonin | 1.040 (62.98) | 0.937 (65.42) | 1.000 (66.24) | 0.950 (62.39)

ADVERSE EVENTS:
Time Frame: From week 0 to week 79 Results are based on the safety analysis set which included all participants who received at least one dose of randomised treatment.
Description: All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during on-treatment period. On-treatment period: the period starting on the date of first administration of trial product and ending on the date of the last dose of trial product +7 days; except for the evaluation of AEs and hypoglycaemic episodes for which the period ended on the date of whatever came first: 1) last dose of trial product + 49 days (7 half lives of semaglutide); 2) end of the in-trial period.
Arm/Group | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/78 | 0/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 12/80 | 15/78 | 12/81 | 8/80
Other Adverse Events (participants affected / at risk) | 61/80 | 64/78 | 63/81 | 55/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.1 mg (N=80) | Semaglutide 0.2 mg (N=78) | Semaglutide 0.4 mg (N=81) | Placebo (N=80)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Transient epileptic amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.1 mg (N=80) | Semaglutide 0.2 mg (N=78) | Semaglutide 0.4 mg (N=81) | Placebo (N=80)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 8 (9) | 4 (7) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 8 (9) | 6 (7) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 6 (7) | 8 (10) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 8 (8) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 5 (5) | 10 (10) | 6 (6)
Constipation (Gastrointestinal disorders) | 12 (14) | 17 (22) | 18 (20) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18) | 18 (18) | 18 (22) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 23 (31) | 22 (30) | 16 (21) | 11 (16)
Dizziness (Nervous system disorders) | 6 (8) | 6 (8) | 8 (10) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 9 (11) | 4 (5) | 5 (7)
Eructation (Gastrointestinal disorders) | 5 (6) | 6 (6) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 8 (8) | 7 (8) | 7 (7)
Flatulence (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 4 (5) | 5 (6) | 2 (2)
Headache (Nervous system disorders) | 7 (11) | 10 (13) | 10 (13) | 8 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (6) | 7 (8)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 3 (3) | 4 (4)
Influenza (Infections and infestations) | 7 (7) | 1 (1) | 3 (4) | 6 (6)
Injection site bruising (General disorders) | 1 (1) | 5 (10) | 3 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (5) | 5 (5)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 4 (5) | 7 (8) | 1 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (15) | 15 (21) | 10 (11) | 12 (22)
Nausea (Gastrointestinal disorders) | 24 (32) | 29 (39) | 33 (49) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (7)
Procedural pain (Injury, poisoning and procedural complications) | 6 (7) | 2 (2) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Sinusitis (Infections and infestations) | 4 (4) | 7 (8) | 2 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (8) | 3 (4) | 5 (6)
Urinary tract infection (Infections and infestations) | 5 (7) | 2 (2) | 7 (9) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (21) | 17 (26) | 12 (29) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02970942/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02970942/SAP_001.pdf